CLINICAL TRIAL: NCT00095927
Title: Phase II, Randomized Study of Concomitant Chemoradiation Using Weekly Carboplatinum/Paclitaxel With (Arm A) or Without (Arm B) Daily Subcutaneous Amifostine in Patients With Newly Diagnosed Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Randomized Amifostine For SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); MedImmune LLC (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Haddad, Robert I.,M.D., Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03018; P30CA006516 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Chemotherapeutic Agent Toxicity; Head and Neck Cancer; Mucositis; Radiation Toxicity; Xerostomia
Keywords: radiation toxicity; chemotherapeutic agent toxicity; mucositis; xerostomia; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Radiation Injuries; Xerostomia; Squamous Cell Carcinoma of Head and Neck | interventions — Amifostine; Carboplatin; Paclitaxel; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A Amifostine (Active Comparator): Patients with newly diagnosed, locally advanced stage ill or IV SCCHN received;
  * 4 weekly doses of carboplatin (area under the curve, 1.5) and paclitaxel (45 mg/m 2) concurrently with concomitant boost radiation consisting of 72 grays in 42 fractions over 6 weeks (every day for 18 days, twice a day for 12 days) (grading determined according to the TNM staging system).
  * Subcutaneous daily amifostine at a dose of 500 mg
  Interventions: Drug: Amifostine; Drug: Carboplatin; Drug: Paclitaxel; Radiation: radiation
- Arm B No-Amifostine (Experimental): Patients with newly diagnosed, locally advanced stage ill or IV SCCHN
  - 4 weekly doses of carboplatin (area under the curve, 1.5) and paclitaxel (45 mg/m 2) concurrently with concomitant boost radiation consisting of 72 grays in 42 fractions over 6 weeks (every day for 18 days, twice a day for 12 days) (grading determined according to the TNM staging system).
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: radiation

INTERVENTIONS:
Drug: Amifostine — Given subcutaneously
  Other Names: Ethyo
  Arms: Arm A Amifostine
Drug: Carboplatin — Given IV
  Other Names: Paraplatin
Drug: Paclitaxel — Given IV
  Other Names: Taxol; Onxal
Radiation: radiation — Given once daily for 4 weeks and then twice daily for 2 weeks.

SUMMARY:
This research study is studying a drug called Amifostine as a treatment for squamous cell carcinoma in the head and/or neck area.

DETAILED DESCRIPTION:
Amifostine is a drug that is used to treat moderate to severe xerostomia (dry mouth) for those who receive radiation therapy for head and neck cancer. It was approved by the FDA for use intravenously. This study plans to examine the effects of xerostomia when Amifostine is used subcutaneously (by injection). Amifostine has been seen to be effective when used to combat the effects of dry mouth, but also has some side effects which are listed later in this consent form.

The purpose of this study is to examine the effectiveness of twice a day radiation therapy given with chemotherapy consisting of carboplatin and paclitaxel (Taxo 1). This study will examine the effectiveness of adding Amifostine in the hopes of reducing the side effects of radiation.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically proven squamous cell carcinoma of the head and neck. Biopsy is preferred unless medically contraindicated.
* Primary tumor sites eligible: oral cavity, oropharynx, hypopharynx or larynx. Tumors of the nasal and paranasal cavities will also be included. Unknown primary SCC in the neck will also be eligible.
* Stage 2, 3 or 4 disease without evidence of distant metastases verified by chest X-Ray, abdominal ultrasound or CT (in case of liver function test abnormalities); bone scan in case of local symptoms.
* At least one uni- or bidimensionally measurable lesion at the start of all therapy (induction therapy ag well as chemoradiation).
* No previous head and neck radiotherapy and no previous curative surgery for SCCHN (other than biopsy) are allowed at time of study entry.
* Age ≥ 18 years.
* WHO performance status of 0 or 1 (section 13, Appendix I)
* No active alcohol addiction (as assessed by medical caregiver).
* Life expectancy ≥ 12 weeks.
* Signed informed consent prior to beginning protocol specific procedures.
* Adequate bone marrow, hepatic and renal functions as evidenced by the following:

  * Hematology:

    * neutrophil count ≥ 2.0 x 10 9/1.
    * platelet count ≥ 100 x 10 9/1.
    * hemoglobin ≥ 10 g/dl.
  * Hepatic function:

    * total bilinthin WNL.
    * ASAT (SGOT) and ALAT (SGPT) ≤ 2.5 x 1JLN.
    * alkaline phosphatase ≤ 5 x ULN.
    * patients with ASAT or ALAT > 1.5 x ULN associated with alkaline phosphatase > 2.5
    * x ULN are not eligible for the study.
  * Renal function: the creatinine clearance ≥ 60 ml/min (actual or calculated by the Cockcroft-Gault method as follows:

    * Weight(kg) x (140 - age)/K x serum creatinine
    * serum creatinine in mg/dL

      * K: 72 in man
      * K: 85 in woman
    * serum creatinine in µmon/L

      * K: 0.814 in man
      * K: 0.96 in woman
* Patients must be available for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centers
* Previous chemotherapy is permitted, provided that it is in induction form before starting radiation therapy and that it is being used to treat head and neck cancers.

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing potential not using adequate contraception.
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin or other cancer curatively treated by surgery and with no evidence of disease for at least 3 years.
* Symptomatic peripheral neuropathy ≥ grade 2 by NCIC-CTG criteria.
* Other serious illnesses or medical conditions including but not limited to:

  * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
  * History of significant neurologic or psychiatric disorders including dementia or seizures.
  * Active uncontrolled infection.
  * Active peptic ulcer.
  * Hypercalcemia.
  * Chronic obstructive pulmonary disease requiring hospitalization during the year preceding study entry.
* Patients requiring intravenous alimentation.
* Patients who experienced a weight loss of more than 20% of their body weight in the 3 months preceding study entry (unless purposeful)
* Concurrent treatment with any other anticancer therapy.
* Participation in an investigational trial within 30 days of study entry.
* Previous treatment with any biologic therapy is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-05; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Rate of local/regional control (LRC) 1 year after beginning treatment | One year after beginning of treatment
Proportion of patients with grade 2 or 3 chronic xerostomia at 3, 6 months | 3, 6 Months
Proportion of patients with grade 3 and 4 mucositis as assessed by RTOG criteria once weekly during and after completion of radiotherapy | End of Radiotherapy
Median duration of dependence on percutaneous endoscopic gastrectomy (PEG) for adequate nutrition at 8, 12, 24, and 52 weeks after completion of study treatment | 8,12, 24 and 52 weeks

SECONDARY OUTCOMES:
Duration of grade 3 and 4 mucositis once weekly during treatment and at 8, 12, 24, and 52 weeks after completion of study treatment | 8, 12, 24, and 52 weeks
Proportion of patients with PEG dependency | 3, 6, and 12 months after completion of study treatment
Time to disease progression | baseline to disease progression
  Kaplan and Meier
Quality of life as assessed by Functional Assessment of Cancer Therapy for Head and Neck Cancer (FACT-H&N) Survey | baseline, 8, 12, 24, and 52 weeks after completion of study treatment
LRC and overall survival at 2 years after completion of study treatment | 2 Years after completion of study treatment
Swallowing function | 2 years Post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert I. Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - Goodall Hospital, Sanford, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Bethke Cancer Center at Emerson Hospital, Concord, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Wentworth Douglass Hospital, Dover, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haddad R, Sonis S, Posner M, Wirth L, Costello R, Braschayko P, Allen A, Mahadevan A, Flynn J, Burke E, Li Y, Tishler RB. Randomized phase 2 study of concomitant chemoradiotherapy using weekly carboplatin/paclitaxel with or without daily subcutaneous amifostine in patients with locally advanced head and neck cancer. Cancer. 2009 Oct 1;115(19):4514-23. doi: 10.1002/cncr.24525. PMID 19634161